CLINICAL TRIAL: NCT06983600
Title: The Effect of SuJok Application on Dysmenorrhea and Quality of Life in Young People With Primary Dysmenorrhea: A Randomized Controlled Study
Brief Title: The Effect of SuJok Application on Dysmenorrhea and Quality of Life in Young People With Primary Dysmenorrhea:
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Collaborators: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, aycan şahin, research assistant, Muş Alparslan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 149972
Record Dates: First submitted 2025-04-03; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Dysmenorrhea (Disorder); Alternative Treatment
Keywords: alternative treatment; primary dysmenorrhea, quality of life
MeSH Terms: conditions — Dysmenorrhea

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): The female students in the study group will be pre-tested by the researcher during the 1st menstrual period before the application. Then, starting from the 1st day of the 2nd month menstrual period for a total of 10 days, the points will be sensitized and the painful point will be detected by the researcher with the macro bug in the hand and the ring in the mini system and the spiral in the hand. Then, moxa will be applied to the reflection point of the uterus and ovary for 2 minutes to 5 minutes. After the moxa application, the black pepper seed will be fixed to the painful point with the help of an airtight plaster. The black pepper seed will be kept for at least 4 hours and maximum 8-10 hours.
  Interventions: Other: alternative therapy:sujok therapy
- Control Arm (No Intervention): In the control group, no application was made during and after the menstrual period.

INTERVENTIONS:
Other: alternative therapy:sujok therapy — As of the first day of the menstrual period for a total of 10 days, the researcher will provide sensitization of the points and painful point detection with the ring and in-hand spiral in the hand macro insect and mini system. Then, moxa will be applied to the uterus and ovary reflection point between 2 minutes and 5 minutes. Moxa is a method that burns wormwood and treats it with the heat emitted to the skin by the smoke with perforated apparatus. It is one of the oldest treatment methods based on heat and plant healing. After the Moxa application, the black pepper seed will be fixed to the painful spot with the help of an air-tight plaster. The black pepper seed will be kept for at least 4 hours and maximum 8-10 hours.
  Arms: Intervention Arm

SUMMARY:
Menarche, which is one of the most prominent features of maturation in adolescents and the transition from childhood to adulthood, causes many problems. The most prominent of these complaints is dysmenorrhea. Primary dysmenorrhea, the most common form of dysmenorrhea, is a gynecological disorder characterized by pain that starts in the lower abdomen before or during menstruation and radiates to the waist and legs.

Primary dysmenorrhea is seen especially in women under 25 years of age and within 6-12 months after menarche. Dysmenorrhea is a preventable and treatable disease. There are pharmacologic and nonpharmacologic methods in the treatment of dysmenorrhea. Pharmacologic methods include NSAIDs and hormonal contraceptives. Nonpharmacological methods used in the treatment of dysmenorrhea include hot application, regulation of nutrition, relaxation exercises, massage, yoga, reflexology, acupuncture, acupressure, TENS method, vitamins B and E, calcium, magnesium, zinc supplements, fennel and rose teas, ginger, aromotherapy applications. In addition to pharmacological methods, nonpharmacological methods are frequently used in the treatment of dysmeorrhea. People have recently turned to alternative medicine in the treatment of diseases in order to get rid of the side effects of drugs. Today, medicine is constantly developing and new treatment options are emerging. The treatment method that has recently started to be used and its effect has been seen is SuJok therapy. SuJok therapy was developed in 1986 by South Korean scientist Professor Park Jae Woo. In Korean, "Su" means hand and "Jok" means foot. In SuJok therapy, hands and feet are used as a treatment method. In SuJok, the hands and feet are a miniature replica of the body and have maximum structural similarity to the human body in anatomical terms. Every organ in our body has reflection points on the hands and feet. Thus, it activates all organs in our body with hands and feet. With the SuJok therapy method, it is argued that by using various techniques with the reflections of the body in the hand and foot points of the body, the organ and body area are physically stimulated and the energy in the body is activated and healing occurs. In the literature, studies on SuJok therapy applications are limited and there are no studies showing the effect of SuJok application on primary dysmenorrhea.

DETAILED DESCRIPTION:
Menarche, which is one of the most prominent features of maturation in adolescents and the transition from childhood to adulthood, also causes many problems. The most prominent of these complaints is dysmenorrhea. Primary dysmenorrhea, the most common form of dysmenorrhea, is a gynecological disorder characterized by pain that starts in the lower abdomen before or during menstruation and radiates to the waist and legs. Although the cause of dysmenorrhea is not clearly known, it is closely associated with menstrual age, prolonged and heavy menstrual blood flow, not having given birth, not being married, body mass index less than 20, eating problems, smoking, presence of chronic disease, physical activity status, low economic status, stress, hirsutism, polycystic ovary syndrome and infertility. In dysmenorrhea, in addition to pain, head, back and leg pain, nausea, vomiting and diarrhea complaints can be seen. During the school period, dysmenorrhea may affect women's academic performance, school attendance, participation in sports activities and social relations with friends.

Primary dysmenorrhea is seen especially in women under 25 years of age and within 6-12 months after menarche. With the first menstruation, progesterone release is low due to corpus luteum insufficiency or more than half of the menstrual cycles are anovulatory. For this reason, dysmenorrhea is seen in cycles with sufficient ovulatory occurrence several menstrual cycles after menarche.

While the prevalence of dysmenorrhea is between 56.2-91.5% in the world, while in our country it is in the range of (66.2- 98.0%).

Dysmenorrhea is a preventable and treatable disease. There are pharmacologic and nonpharmacologic methods in the treatment of dysmenorrhea. Pharmacologic methods include NSAIDs and hormonal contraceptives. Nonpharmacological methods used in the treatment of dysmenorrhea include hot application, regulation of nutrition, relaxation exercises, massage, yoga, reflexology, acupuncture, acupressure, TENS method, vitamins B and E, calcium, magnesium, zinc supplements, fennel and rose teas, ginger, aromotherapy applications. In addition to pharmacological methods, nonpharmacological methods are frequently used in the treatment of dysmeorrhea. People have recently turned to alternative medicine in the treatment of diseases in order to get rid of the side effects of drugs. Today, medicine is constantly developing and new treatment options are emerging. The treatment method that has recently started to be used and its effect has been seen is SuJok therapy. SuJok therapy was developed in 1986 by South Korean scientist Professor Park Jae Woo. In Korean, "Su" means hand and "Jok" means foot. In SuJok therapy, hands and feet are used as a treatment method. In SuJok, the hands and feet are a miniature replica of the body and have maximum structural similarity to the human body in anatomical terms.

Every organ in our body has reflection points on the hands and feet. Thus, it activates all organs in our body with hands and feet. With the SuJok therapy method, it is argued that by using various techniques with the reflections of the body in the hand and foot points of the body, the organ and body area are physically stimulated and the energy in the body is activated and healing occurs. Studies on SuJok therapy applications are limited in the literature and there are no studies showing the effect of SuJok application on primary dysmenorrhea.

In order to determine the effects on the fear levels experienced by patients diagnosed with Covid-19, it was determined that insemination with bending as SuJok therapy application significantly reduced the fear levels. In the study conducted by Pérez Cruz et al., it was determined that the Su Jok therapy application applied to 30 people with cervical pain decreased significantly compared to those in the control group. They found that there was a significant difference in the 60th minute of seed application to 24 migraine patients with SuJok therapy compared to the control group. The advantages of SuJok application are that it is easy to apply, has no side effects, does not involve an interventional application and has a large surface area as application sites.

The research will be conducted to determine the effect of sujok therapy on dysmenorrhea and quality of life in young people with primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:- Being a female student studying in the 1st or 2nd year at the Faculty of Health Sciences,

* Scoring menstrual pain 5 and above out of 10 points on the VAS Visual Pain Scale,
* Don't be nullipar,
* Regular mentruation for at least the last six months,
* Not having any gynecological diagnosis,
* Not having undergone any gynecological operation,
* Willingness and acceptance to participate in the study,
* In addition, students who do not have any lesions, infections, etc. that prevent the application of water jok therapy on the hands and feet

Exclusion Criteria:

* - Scoring 4 or less out of 10 points on the VAS Visual Pain Scale,
* Participants who volunteered to participate in the study and wanted to leave at any stage

Ages: 18 Months to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Pre and Post Intervention Dysmenorrhea Follow-up Form | Pain intensity reported at baseline, day 1 and day 10 of menstruation after intervention
  1. In the first part, the premenstrual dysmenorrhea follow-up form is applied. The pain felt in the form is evaluated using the Visual Analog Scale (VAS). 0-10; 0- No pain, 10- Worst pain.
World Health Organization Quality of Life Scale-Short Form (WHOQOL-BREF) | Pain intensity reported at baseline, day 1 and day 10 of menstruation after intervention
  WHOQOL-BREF is a valid and reliable scale developed by the World Health Organization to assess health-related quality of life. The short form of the scale includes 27 questions. These questions give physical, mental, social and environmental scores. The score that each area can get independently of each other is between 4-20. The increase in the score indicates an increase in quality of life.
Dysmenorrhea Follow-up Form after Sujok therapy application | Pain intensity reported at baseline, day 1 and day 10 of menstruation after intervention
  After the su jok therapy applied during menstruation, a dysmenorrhea follow-up form is applied. The pain felt in the form is evaluated using the Visual Analog Scale (VAS). 0-10; 0- No pain, 10- The worst pain.

CONTACTS AND LOCATIONS:
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
It was planned to share basic information such as the age, education level, place of residence, smoking status, height-weight ratio, knowledge about menstruation, how long menstrual pain lasts, whether there is a relative in the family who has pain during menstruation, whether they use painkillers, if so, who recommended them, whether they do anything other than painkillers to relieve menstrual pain, and if so, what they are, whether your menstrual pain affects your daily activities and school attendance. Basic comparison results with the World Health Organization Quality of Life Scale-Short Form (WHOQOL-BREF) and Visual Assessment Scale (VAS) scales will be shared.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The study is planned to be finalized from April 2025 to September 2025. the translation of the results into an article is planned to be done until December 2025.
Access Criteria: For variables with two groups, the independent groups t-test and the non-parametric Mann Whitney U test, and for variables with at least three or more groups, the one-way analysis of variance and the non-parametric Kruskall Wallis H test were considered.
  In the analysis of the differences and changes between two measurements over time in groups, the t-test was used in dependent groups in groups that met the assumption of normal distribution, and the Wilcoxon signed-rank test was used in groups that did not meet the assumption of normal distribution. Again, in the analysis of the differences and changes between three or more measurements according to time in the groups, it was planned to use one-way analysis of variance in repeated measures in groups that meet the assumption of normal distribution, and Friedman test in groups that do not meet the assumption of normal distribution. Statistical significance level will be accepted as p<0.05 in all tests.